CLINICAL TRIAL: NCT01857440
Title: The Flashing Light-Induced Pupil Response (FLIPR) Glaucoma Study
Acronym: FLIPR
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Andrew Hartwick, Assistant Professor, Ohio State University
Other Study IDs: 2013H0073; 8KL2TR000112-05 (NIH)
Record Dates: First submitted 2013-05-13; First posted 2013-05-20 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Glaucoma, Open-Angle; Eye Diseases
Keywords: Glaucoma; Pupil; Melanopsin
MeSH Terms: conditions — Glaucoma, Open-Angle; Eye Diseases; Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects with glaucoma (Cases): This group will consist of patients with glaucoma who are under care at the Ohio State University Havener Eye Institute.
- Subjects without glaucoma (Controls): This group will consist of matched controls who are free of glaucoma and other complications, and who received a comprehensive eye examination at the Ohio State University College of Optometry.

SUMMARY:
This study is designed to investigate whether the pupil response to slowly flashing colored lights is significantly altered in patients with glaucoma, as compared to a control group of subjects without glaucoma.

DETAILED DESCRIPTION:
The pupils inside the eyes constrict in response to light stimulation. Different classes of cells within the human retina initiate this response. Recent research suggests that one of the ganglion cell types involved in this pupil response is affected by glaucoma. By measuring pupil responses to different colored lights, the function of this class of cells can be evaluated quickly, and without touching the eye. An advantage of pupil testing strategies is that they do not require subjective feedback from the subject about what they can see, as is required for standard visual field tests that are used in the clinic.

The main aim of this study is to measure and compare the pupil constriction that occurs in response to flickering red and blue lights in patients with glaucoma versus matched control patients without glaucoma. In addition, the subjects will be asked questions about their quality of life and it will be determined whether issues related to quality of life correlate to alterations in the pupil responses.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Diagnosed with glaucoma of known severity (cases only)
* Have a refractive error between +4.00 and -8.00 sphere power, and no more than 3.00 diopters of astigmatism
* Best corrected visual acuity of 20/40 or better in each eye
* Have open anterior chamber angles

Exclusion Criteria:

* Diagnosis of glaucoma of a type other than Primary Open Angle (cases only)
* History of having surgery or taking medications known to profoundly affect pupillary function or shape
* Visual Field defect (controls only)
* History of traumatic brain injury requiring hospitalization
* Pregnancy
* History of optic nerve disease other than glaucoma
* History of retinopathy
* History of unreactive pupils
* Presence of significant cataract

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases: Age 18 or older with diagnosed glaucoma of known severity Controls: Matched to Cases on age, sex, and race.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pupil Response | Single Visit: One Day
  Using fourier analysis, the pupil fluctuation evoked by blue and red flickering lights will be measured in glaucoma patients and compared to matched controls.

SECONDARY OUTCOMES:
Quality of Life Survey | Single Visit: One Day
  Subjects will fill out a questionnaire with questions that assess quality of life issues, and the results will be correlated to the pupil response data.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hartwick, OD, PhD, Principal Investigator — OSU College of Optometry
Locations (2):
- United States (2):
  - OSU College of Optometry, Columbus, Ohio
  - Havener Eye Institute, Columbus, Ohio

REFERENCES:
- [Result] Shorter P, Eren D, Jain SG, Hartwick ATE. 2014. The flashing light-induced pupil response (FLIPR) glaucoma study. Invest. Ophthalmol. & Vis. Sci. 55: E-abstract 5608.